CLINICAL TRIAL: NCT06037395
Title: A Randomized, Double-blind, Two-arm, Parallel Group, Single-dose, Phase I Study to Compare the Pharmacokinetics, Pharmacodynamics, and Safety Between CT-P41 and US-licensed Prolia in Healthy Male Subjects
Brief Title: Phase I Study to Compare the Pharmacokinetics, Pharmacodynamics, and Safety Between CT-P41 and US-licensed Prolia in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-P41 1.2
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Healthy Subject
Keywords: CT-P41

STUDY DESIGN:
Intervention Model Description: Two-arm, Parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT-P41 (Experimental): a single 60 mg subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P41
- US-licensed Prolia (Active Comparator): a single 60 mg subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: US-licensed Prolia

INTERVENTIONS:
Biological: CT-P41 — a single 60 mg subcutaneous (SC) injection via pre-filled syringe (PFS)
  Arms: CT-P41
Biological: US-licensed Prolia — a single 60 mg subcutaneous (SC) injection via pre-filled syringe (PFS)
  Arms: US-licensed Prolia

SUMMARY:
A Randomized, Double-blind, Two-arm, Parallel group, Single-dose, Phase I Study to Compare the Pharmacokinetics, Pharmacodynamics, and Safety between CT-P41 and US-licensed Prolia in Healthy Male Subjects

DETAILED DESCRIPTION:
This study was a randomized, double-blind, two-arm, parallel group, single-dose, phase I study designed to compare PK, PD, safety, and immunogenicity between CT-P41 and US-licensed Prolia in healthy male subjects. Subjects were randomized into a 1:1 ratio to receive a single dose (60 mg) of either CT-P41 or US-licensed Prolia. The subjects were followed up for 253 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, between the ages of 28 and 55 years, both inclusive
2. Subject had a body mass index (BMI) between 18.5 and 29.9 kg/m2, both inclusive, and a body weight between 50.0 and 99.9 kg, both inclusive, when rounded to the nearest tenth.
3. Subject with total serum calcium ≥ 8.5 mg/dL (≥ 2.125 mmol/L) and serum 25-OH vitamin D ≥ 20 ng/mL (≥ 50 nmol/L)

Exclusion Criteria:

1. Subject was a female.
2. Subject with a hypersensitivity to any component of denosumab or dry natural rubber (a derivative of latex).
3. Subject was confirmed or suspected with infection of coronavirus disease 2019 (COVID-19) at screening, or had had contact with COVID-19 patient within 14 days from screening.
4. Subject had a medical history of and/or current medical condition that can have effect on the study. Details to be discussed with investigator as per Protocol.

   1. Subjects with known risk factors for hypocalcaemia
   2. Subjects with known intolerance to calcium or vitamin D supplements
   3. Subjects with known infection with active hepatitis B, hepatitis C, human immunodeficiency virus, or syphilis
5. Subject had a history of and/or concurrent use of medications including any prior therapy that can have effect on the study. Details to be discussed with investigator as per Protocol.
6. Subjects have or had any therapy that might significantly affect bone metabolism

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
AUCinf | up to Day 253
  Area under the concentration-time curve from time zero to infinity (AUC0-inf)
AUClast | up to Day 253
  Area under the concentration-time curve from time zero to the last quantifiable concentration (AUC0-last)
Cmax | up to Day 253
  maximum serum concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - CHA Bundang Medical Center, Seongnam, Bundang-gu
  - Chungnam National University Hospital, Daejeon, Jung-gu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim A, Hong JH, Shin W, Yoo H, Jung JG, Reginster JY, Kim S, Bae Y, Suh J, Kim S, Lee E, Silverman S. A randomized, double-blind, single-dose, phase 1 study comparing the pharmacokinetics, pharmacodynamics, safety, and immunogenicity of denosumab biosimilar CT-P41 and reference denosumab in healthy males. Expert Opin Biol Ther. 2024 Jul;24(7):655-663. doi: 10.1080/14712598.2024.2316846. Epub 2024 Feb 22. PMID 38349618